CLINICAL TRIAL: NCT06997835
Title: Research on the Preventive Effect of Family-centered Early Nursing Intervention on High-risk Population of Gestational Diabetes Mellitus
Brief Title: The Role of Early Nursing Intervention in the High-risk Population of Gestational Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yan Lu (Other)
Responsible Party: Sponsor-Investigator, Yan Lu, Clinical Professor, Nantong First People's Hospital
Organization: Nantong First People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025XM105
Record Dates: First submitted 2025-05-14; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Early Nursing Intervention; Gestational Diabetes Mellitus
Keywords: Gestational diabetes mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental)
  Interventions: Behavioral: Control group：The interactive management nursing model on the wechat platform
- Intervention group (Experimental)
  Interventions: Behavioral: Intervention group：Family-centered early care intervention

INTERVENTIONS:
Behavioral: Control group：The interactive management nursing model on the wechat platform — The intervention subjects of the control group: targeted at the pregnant and postpartum women themselves. Specifically, conduct routine outpatient prenatal examinations and health education for pregnant women. Regularly receive health education and pregnancy guidance intervention provided by the wechat platform. It includes: ① Setting specific wechat ringtones, 60-second voice messages and picture reminders every day; ② Basic knowledge education every Monday ③ Dietary guidance is provided every Tuesday. ④ Exercise guidance every Wednesday ⑤ Guidance on blood glucose monitoring every Thursday; Weight guidance is provided every Friday.
  Arms: Control group
Behavioral: Intervention group：Family-centered early care intervention — The intervention subjects of the intervention group were parturients and their primary caregivers (spouses and parents).
  The specific measures are as follows:
  1. Establish a family-centered healthcare team (FCC) It includes one chief physician, two attending physicians, one diabetes specialist nurse, two responsible nurses, one psychotherapist, and one nutritionist. The organization members will conduct FCC concept learning and knowledge training.
  2. Interactive management nursing model on the wechat platform
     * Set specific wechat ringtones, 60-second voice messages and picture reminders every day;
       * Basic knowledge education every Monday; ③. Dietary guidance every Tuesday;
         ④. Exercise guidance every Wednesday;
         ⑤ Guidance on blood glucose monitoring every Thursday;
         ⑥. Weight guidance every Friday;
         ⑦. Strengthen home care guidance every Saturday and Sunday.
  Arms: Intervention group

SUMMARY:
Pregnant women who established prenatal examination cards in the prenatal outpatient department of our hospital from January 2025 to September 2025 were selected. According to the inclusion criteria, 200 high-risk pregnant women with gestational diabetes mellitus (GDM) were selected. 100 people in the control group received conventional nursing intervention measures, and 100 people in the intervention group adopted the family-centered wechat platform interactive management nursing model. The observation period was from the start of prenatal examination to follow-up until delivery. The blood glucose conditions, glycated hemoglobin (HbA1c) levels, incidence of GDM, and weight gain during pregnancy of the two groups of pregnant women were observed. The pregnancy outcomes included: Gestational age at delivery, gestational complications (gestational hypertension, diabetic ketosis, preterm birth, post-term pregnancy, urogenital tract infection), polyhydramnios, mode of delivery (induced labor, shoulder dystocia, cesarean section), premature rupture of membranes, postpartum complications (postpartum hemorrhage, puerperal infection), etc. Perinatal outcomes: including fetal growth restriction, macrosomia, preterm birth, stillbirth, fetal malformations, fetal distress, neonatal respiratory distress syndrome, neonatal hypoglycemia, etc. We applied FCC to pregnant women at high risk of gestational diabetes mellitus (GDM) and advanced the intervention window to the beginning of prenatal examination (8-10 weeks of pregnancy). This may be able to improve weight gain and blood glucose levels during pregnancy in high-risk pregnant women, reduce the incidence of GDM, improve the final maternal and infant outcomes, and provide a certain theoretical basis for prenatal nursing intervention in pregnant women at high risk of GDM in the future.

ELIGIBILITY:
Inclusion Criteria:

Gestational age <10 weeks Singleton pregnancy confirmed by first-trimester ultrasound

Primary caregiver availability: At least one primary caregiver (spouse or parent) who:

1. Demonstrates adequate verbal communication and literacy skills (assessed by standardized evaluation)
2. Voluntarily participates in the study with signed informed consent

Metabolic risk factors meeting ≥1 criterion:

1. Pre-pregnancy BMI >24 kg/m²
2. Maternal age ≥35 years at conception
3. Documented history of polycystic ovary syndrome (PCOS)
4. Fasting blood glucose (FBG) ≥5.1 mmol/L in early pregnancy
5. Parental history of diabetes mellitus (either parent)
6. Previous gestational diabetes mellitus (GDM)
7. History of macrosomia (birth weight ≥4000g)
8. Adverse obstetric history including:

Preterm delivery (<37 weeks) Stillbirth or fetal demise Congenital malformations Neonatal death or unexplained neonatal death

Exclusion Criteria:

Pre-existing medical conditions:

1. Chronic hypertension (diagnosed pre-pregnancy)
2. Renal disorders (e.g., chronic kidney disease stage ≥3)
3. Cardiovascular diseases (e.g., coronary artery disease, heart failure)

Prohibited medication use during pregnancy including:

1. Indomethacin
2. Phentolamine
3. Diuretics (e.g., furosemide, hydrochlorothiazide)
4. Phenytoin
5. Systemic corticosteroids (e.g., cortisone, prednisone)

Activity-limiting comorbidities:

a) Severe medical complications contraindicating physical activity (e.g., unstable angina, advanced respiratory failure)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of gestational diabetes | 24 weeks of gestation
  The number of cases of GDM/the total number of observed cases

SECONDARY OUTCOMES:
Blood sugar status of pregnant women | 24 weeks of gestation
  The occurrence of abnormal OGTT (OGTT examination was performed at 24 weeks, and fasting, 1-hour, and 2-hour blood glucose were measured), and the level of glycated hemoglobin (HbA1c)
The weight gain of pregnant women during pregnancy | From randomization to pregnancy termination (maximum assessment time: 42 weeks of gestation)
  The pre-pregnancy BMI was lower than the normal value, and the weight gain during pregnancy was 12.5-18.0kg. Those with a normal BMI before pregnancy gained 11.5 to 16.0kg during pregnancy. Those with an excessive BMI before pregnancy gained 7.0 to 11.5 kilograms during pregnancy. Obese people before pregnancy gain 5.0 to 9.0 kilograms during pregnancy. Weight gain during pregnancy is classified into three levels: insufficient weight gain, appropriate weight gain, and excessive weight gain. If the weight gain during pregnancy is less than the corresponding pre-pregnancy BMI weight gain range, it is considered insufficient weight gain; if it is greater than the corresponding weight gain range, it is considered excessive weight gain.
Gestational weeks at delivery | From pregnancy confirmation to delivery (range: ≥20 weeks to ≤42 weeks)
  Gestational age at delivery (based on the gestational age confirmed by the last menstrual period or early ultrasound)
Complications during pregnancy | From enrollment to delivery
  Clinical diagnosis of gestational hypertension, preeclampsia, diabetic ketoacidosis, preterm birth (<37 weeks), post-term pregnancy (≥42 weeks), and urogenital tract infections
Polyhydramnios | Middle and late stages of pregnancy (such as being evaluated every 4 weeks after 20 weeks of pregnancy until delivery)
  Ultrasound diagnosis: Amniotic fluid index (AFI) >24 cm or maximum vertical amniotic fluid depth (MVP) >8 cm
Postpartum complications | From delivery to discharge (or within 42 days after delivery)
  The incidence of postpartum hemorrhage (blood loss ≥500ml) and puerperal infection (body temperature ≥38℃+ laboratory confirmation)
Mode of delivery | Records during childbirth
  The incidence rates of induced labor, shoulder dystocia and cesarean section
Premature rupture of membranes | Pregnancy ≥37 weeks until before delivery
  Clinical diagnosis of natural rupture of membranes before labor
The length and cost of hospital stay after delivery | From delivery to discharge
  Length of hospital stay (days) and total cost
Fetal growth restriction | The assessment should be conducted every 4 weeks after 20 weeks of pregnancy until delivery
  Ultrasound assessment of fetal weight < the 10th percentile at the same gestational week
Macrosomia | Records during childbirth
  Birth weight ≥4000g
Premature birth | From enrollment to delivery
  The gestational age at delivery is less than 37 weeks
Stillbirth | From enrollment to delivery
  Fetal death occurs after ≥20 weeks of pregnancy
Fetal malformation | During the second trimester of pregnancy (18-24 weeks) and within 24 hours after birth
  Congenital malformations confirmed by ultrasound or clinically after birth
Fetal distress | Records during childbirth
  Abnormal fetal heart rate monitoring (such as repeated late deceleration) or amniotic fluid fecal contamination
Neonatal respiratory distress syndrome | Within 7 days after birth
  Clinical diagnosis (aerobic therapy or ventilator support + chest X-ray confirmation)
Neonatal hypoglycemia | Within 24 hours after birth
  Blood glucose <2.6mmol/L (at least two tests are required for confirmation)
The rate of newborns admitted to the NICU | From birth to discharge (or within 28 days after birth)
  Indications and days of transfer to the Neonatal Intensive Care Unit (NICU)

CONTACTS AND LOCATIONS:
Locations (1):
- Nantong First People's Hospital, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No